CLINICAL TRIAL: NCT00439192
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Phase II, Forced Dose Titration Study to Investigate the Efficacy and Safety of 400mg and 600mg ELB245 Given Once Daily for 12 Weeks (8 + 4 Weeks) Versus Placebo and Versus 4mg Tolterodine Given Once Daily in Patients With Incontinent Overactive Bladder (OAB)
Brief Title: ELB245 for 12 Weeks Versus 4mg Tolterodine in Patients With Incontinent Overactive Bladder (OAB)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: side effect profile did not match expectations
Sponsor: elbion AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELB245201-06
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: OAB, proof of concept; Overactive Bladder (OAB); with incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: ELB245
Drug: Tolterodine

SUMMARY:
This study is designed to determine the efficacy of escalating doses of ELB245 versus placebo , when administered to patients with OAB and to compare the efficacy of escalating doses of ELB245 versus the standard treatment tolterodine, when administered to patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age
* Symptoms of OAB for a minimum of 3 consecutive months prior to study entry; severity of OAB (as defined by patient reported symptoms) for a minimum of one month prior to study entry
* Ability to use a toilet independently and without difficulty
* No treatment with any medication against OAB during the 4 weeks prior to study entry
* Written informed consent

Exclusion Criteria:

* Breastfeeding women, pregnant women or women who intend to become pregnant during the study or women of childbearing potential who are sexually active and not practicing a highly reliable method of birth control
* Any local pathology, that might cause the bladder symptoms
* Significant stress urinary incontinence or mixed stress/urgency incontinence
* Any neurological disease affecting bladder function or muscle strength
* Patient history of any lower urinary tract surgery or previous pelvic irradiation
* Local administration of botulinum toxin within the last 9 months in the lower urinary tract
* Start or change of a behavioral bladder training program
* Post voiding residual volumes larger than 250ml or symptoms of clinically relevant bladder outlet obstruction
* Nocturial polyuria
* History of liver disease and/or impaired liver function
* Cholestasis
* Chronic alcohol or drug abuse
* Evidence of significantly impaired renal function (
* Diabetes mellitus (type I or II) with significant peripheral neuropathy and/or polyuria
* Inflammatory bowel disease such as Crohn's disease, or ulcerative colitis
* Uncontrolled narrow angle glaucoma
* Chronic use of carbamazepine or paracetamol
* Participation in any drug study in the preceding 3 months
* Concomitant treatment with strong CYP3A4 inhibitors
* History or evidence of relevant cardiovascular or cerebrovascular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2007-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
mean number of micturitions

SECONDARY OUTCOMES:
OAB related measures
urgency measures
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Martin Michel, Prof., Study Chair — Dept. Pharmacology & Pharmacotherapy, AMC, University of Amsterdam
Locations (28):
- Germany (15):
  - Private Gynecological Practice, Alzey
  - Private Urologic Practice, Berlin
  - Private Urologic Practice, Borken
  - Private Urologic Practice, Duisburg
  - Private Urologic Practice, Essen
  - Private Urologic Practice, Greifswald
  - Private Urologic Practice, Hamburg
  - Private Urologic Practice, Homburg Saar
  - Private Urologic Practice, Kleinblittersdorf
  - Private Urologic Practice, Marburg
  - Private Urologic Practice, Munich
  - Private Urologic Practice, Mühlacker
  - Private Urologic Practice, Mülheim
  - Private Urologic Practice, Oberursel
  - Private Urologic Practice, Stuttgart
- Poland (9):
  - NZOZ Centrum Medyczne dr n. med. Artur Racewicz, Bialystok
  - Urovita Sp z o.o., Chorzów
  - Invicta Sp z o.o., Gdansk
  - Szpital Specjalistyczny w Koscierzynie, Dep. Oddzial Urologii, Kościerzyna
  - NZOZ Specjalista Sp. z o.o., Kutno
  - NZOZ Nasz Lekarz, Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna, Torun
  - Szpital Kliniczny - Centrum Leczenia Obrazen "Dzieciatka Jezus", Warsaw
  - Centrum Leczenia Chorob Cywilizacyjnych Andrzej Opadczuk, Warsaw
  - EMC Instytut Medyczny S.A., EuroMediCare, Szpital Specjalistyczny z Przychodnia, Wroclaw
- Sweden (4):
  - University Hospital Linköping, Linköping
  - Karolinska University Hospital Huddinge, Stockholm
  - Danderyds Hospital, Stockholm
  - University Hospital Uppsala, Uppsala

REFERENCES:
- [Derived] Song T, Hayanga J, Durham L, Garrison L, McCarthy P, Barksdale A, Smith D, Bartlett R, Jaros M, Nelson P, Molnar Z, Deliargyris E, Moazami N. CytoSorb Therapy in COVID-19 (CTC) Patients Requiring Extracorporeal Membrane Oxygenation: A Multicenter, Retrospective Registry. Front Med (Lausanne). 2021 Dec 20;8:773461. doi: 10.3389/fmed.2021.773461. eCollection 2021. PMID 34988092